CLINICAL TRIAL: NCT00879502
Title: Limbic System Function in Carriers of the Fragile X Premutation
Brief Title: Examining Physiology and Brain Function in People With the Fragile X Premutation
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200614734; R01MH078041 (NIH); DDTR B2-MBA
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Fragile X Premutation
Keywords: Fragile X Premutation; FMR1; Premutation; Fragile X; Brain Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Men with the fragile X premutation
- 2: Healthy men
- 3: Brothers of men with the fragile X premutation

SUMMARY:
This study will examine whether individuals with the fragile X genetic premutation are likely to have emotional, social, and memory deficits and how the brain may be involved in these deficits.

DETAILED DESCRIPTION:
FMR1 is a gene associated with fragile X syndrome-the most common cause of mental retardation-and with social, emotional, and cognitive deficits. The chance of developing these deficits depends on the number of times the FMR1 gene is repeated on the X chromosome. Individuals with more than 200 copies of the FMR1 gene have the full fragile X mutation, putting them at most risk for mental retardation. Individuals with between 55 and 200 copies of the FMR1 gene have the fragile X premutation; they are much less likely to develop mental retardation, but they may have subtle social, emotional, and cognitive deficits and their children are more likely to have the full fragile X mutation. A theory, which this study will test, holds that the deficits of people with the fragile X premutation are caused by dysfunction in the limbic system. The limbic system consists of a group of structures in the brain that govern emotions and behavior. This study will examine people with the fragile X premutation to determine whether and to what extent they have emotional, social, and memory deficits. The study will also determine whether changes in fragile X gene function are related to increased deficits and how the brain, and specifically the limbic system, may be involved in these deficits.

Participation in this study will last 2 days. Participants will undergo several hours of testing at a lab on back-to-back days. Testing on the first day will include the following: providing several saliva samples; undergoing neuropsychological testing, in which participants will solve different types of problems and be interviewed about their emotional and social experiences; and undergoing a physical exam and blood draw.

Testing on the second day will include the following: an MRI scan, which will take pictures of the brain both while participants are resting and while they are performing certain tasks; more neuropsychological testing similar to that from the day before; and questionnaires about emotional and social experiences. A family member will also be asked to fill out a questionnaire about the participant. On 2 other days, participants will be asked to collect saliva samples while at their homes and send the samples to the study researchers. In addition, the researchers will keep in contact with participants in case any follow-up is needed over the next few years.

ELIGIBILITY:
Inclusion Criteria:

* Possesses FMR1 premutation or is part of the general population control group
* Normal or corrected vision
* Speaks English

Exclusion Criteria:

* Presence of contraindication for brain MRI, such as having metal in the body
* Presence of a major medical condition, such as kidney, heart, or liver disease
* Presence of a neurological disorder
* Current alcohol or drug abuse or dependence
* History of head trauma
* History of brain infection
* Medication affecting cerebral blood flow

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Members of the general population, those with the fragile X premutation, and the brothers of those with the fragile X premutation
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2007-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Amygdala and hippocampus volume and function | Age at time of visit

CONTACTS AND LOCATIONS:
Locations (1):
- M.I.N.D. Institute, U.C. Davis, Sacramento, California, United States

REFERENCES:
- See also: Click here for information on the M.I.N.D. Institute — http://www.ucdmc.ucdavis.edu/mindinstitute/